CLINICAL TRIAL: NCT04563026
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2b Study to Evaluate Safety and Efficacy of DUR-928 in Subjects With Alcoholic Hepatitis
Brief Title: A Phase 2b Study in Subjects With Alcoholic Hepatitis to Evaluate Safety and Efficacy of DUR-928 Treatment
Acronym: AHFIRM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Durect (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C928-011
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; acute alcoholic liver disease; progressive inflammatory liver injury
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Intervention Model Description: This is a Phase 2b randomized, double-blind, placebo-controlled, multi-arm, multi-center, parallel design trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DUR-928 (larsucosterol, 30 mg) (Experimental)
  Interventions: Drug: DUR-928 30 mg
- DUR-928 (larsucosterol, 90 mg) (Experimental)
  Interventions: Drug: DUR-928 90 mg
- (Placebo) Sterile Water for Injection (Placebo Comparator)
  Interventions: Drug: Placebo+ Standard of Care (SOC)

INTERVENTIONS:
Drug: DUR-928 30 mg — IV infusion
  Arms: DUR-928 (larsucosterol, 30 mg)
Drug: DUR-928 90 mg — IV infusion
  Arms: DUR-928 (larsucosterol, 90 mg)
Drug: Placebo+ Standard of Care (SOC) — IV infusion
  Arms: (Placebo) Sterile Water for Injection

SUMMARY:
This is a randomized, double-blind, placebo-controlled, phase 2b clinical Trial evaluating Safety and Efficacy of DUR-928 (an experimental medication) in Patients with Alcoholic Hepatitis (AH).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent (either from subject or subject's legally acceptable representative).
2. Onset of jaundice within prior 8 weeks.
3. Average daily consumption of >40 (females) or >60 (males) grams of alcohol for 6 months or longer, with < 8 weeks of abstinence before the onset of jaundice.
4. The determination of AH may be based on typical serum chemistry (as determined by local laboratory) or liver biopsy at any time during the current episode of AH:

   * Serum total bilirubin > 3.0 mg/dL
   * 50 < AST < 400 IU/L
   * ALT < 400 IU/L
   * AST/ALT > 1.5
5. Maddrey discriminant function (MDF) ≥ 32 assuming a control prothrombin time of 12 seconds.
6. Model for End-stage Liver Disease (MELD) score: 21-30.
7. Liver biopsy is not required, but may be used to confirm the diagnosis of AH at the Investigator's discretion. Biopsy, if used as a diagnostic criterion, must have occurred during the current episode.
8. Male or female subjects 18 years of age or older.
9. Subjects must agree to use effective methods to prevent pregnancy while participating in the study.
10. Subjects must agree to participate in an alcohol abstinence support program recommended by the local institution's addiction specialists.

Exclusion Criteria:

1. Subjects taking systemic corticosteroids for a duration exceeding 8 days in the 30 days prior to screening.
2. Subjects experiencing or considered at high risk for alcohol withdrawal seizures or delirium tremens.
3. Active infection (such as spontaneous bacterial peritonitis [SBP], urinary tract infection [UTI], bacteremia, acute viral hepatitis, uncontrolled HIV, and active SARS CoV2 infection).
4. Serum creatinine >2.5 mg/dL.
5. Subjects undergoing continuous veno-venous hemodialysis (CVVH).
6. Uncontrolled gastrointestinal bleeding.
7. A history of pre-admission refractory ascites defined as more than 4 paracenteses in the previous 8 weeks despite diuretic therapy.
8. Liver biopsy (if carried out) with findings not compatible with AH.
9. Stage ≥3 hepatic encephalopathy by West Haven criteria.
10. Any severe concomitant cardiovascular, renal, endocrine, pulmonary, psychiatric disorder, or multi-organ failure.
11. Other concomitant cause(s) of liver disease.
12. Any active malignancy or any malignancy diagnosed within the last five years other than curable skin cancer (basal cell or squamous cell carcinomas).
13. Positive Urine Drug Screen (amphetamines, barbiturates, benzodiazepines, cocaine and opiates) except THC and prescription medications.
14. Existing or intended pregnancy or breast feeding.
15. Participation in another interventional clinical trial within 30 days of Screening.
16. History of organ transplantation, other than a corneal transplant.
17. Underlying diseases that, in the opinion of the site investigator, might be complicated or exacerbated by proposed treatments or might confound assessment of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Difference in 90-day mortality or liver transplant between IV DUR-928, 30 mg or 90 mg, and placebo. | Day 90

SECONDARY OUTCOMES:
Difference in 90-day mortality between IV DUR-928, 30 mg or 90 mg, and placebo. | Day 90
Difference in 28-day mortality or liver transplant between IV DUR-928, 30 mg or 90 mg, and placebo. | Day 28
Difference in 28-day mortality between IV DUR-928, 30 mg or 90 mg, and placebo. | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gordon, MD, FACS, Study Director — CTI Clinical Trial and Consulting Services
Locations (68):
- United States (48):
  - University of Alabama at Birmingham (UAB) Hospital, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Southern California Research Center, Coronado, California
  - Keck Hospital of University of Southern California (USC), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis (UC Davis) Medical Center, Sacramento, California
  - University of California San Francisco (UCSF) Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Health - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Richard Roudebush VA Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Saint Luke's Health System - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center (UNMC), Omaha, Nebraska
  - Rutgers-New Jersey Medical School, Newark, New Jersey
  - University of New Mexico (UNM) Hospital, Albuquerque, New Mexico
  - Northwell Health - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Hospital, New York, New York
  - New York-Presbyterian - Weill Cornell Medical Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina (MUSC) Health - University Medical Center, Charleston, South Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Baylor Scott and White Health, Dallas, Texas
  - University of Texas Southwestern (Clements University Hospital), Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Doctors Hospital at Renaissance (DHR), Edinburg, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Utah Health - The University of Utah Hospital, Salt Lake City, Utah
  - University of Virginia (UVA) Health - University Hospital, Charlottesville, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Harborview Medical Center - University of Washington, Seattle, Washington
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Mater Health - Mater Hospital Brisbane, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Landeskrankenhaus (LKH) - Universitätsklinikum Graz, Graz, Austria
- Belgium (2):
  - Université libre de Bruxelles (ULB) - Hôpital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA), Edegem
- France (4):
  - Centre Hospitalier Régional Universitaire (CHRU) Besançon - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier Universitaire (CHU) de Lille - Hôpital Jeanne de Flandre, Lille
  - Hospices Civils de Lyon - Hôpital de la Croix-Rousse, Lyon
  - Hôpital St Joseph, Marseille
- United Kingdom (5):
  - Barts Health NHS Trust - The Royal London Hospital, London, England
  - King's College Hospital NHS Foundation Trust, London, England
  - Imperial College Healthcare NHS Trust - St. Mary's Hospital, London, England
  - University Hospitals Plymouth NHS Trust - Derriford Hospital, Plymouth, England
  - Royal Free London NHS Foundation Trust Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiffman M, Da B, Goel A, Kwong A, Stein L, Moreno C, Nicoll A, Mehta A, Louvet A, Flamm S, Pyrsopoulos N, Satapathy S, Kuo A, Ganger D, Aloman C, Strasser SI, Tse E, Russo MW, Rockey D, Gray M, Mitchell M, Thursz M, Krebs W, Scott D, Blevins C, Ellis D, Brown J, Sussman N, Lin W. Larsucosterol for the Treatment of Alcohol-Associated Hepatitis. NEJM Evid. 2025 Feb;4(2):EVIDoa2400243. doi: 10.1056/EVIDoa2400243. Epub 2025 Jan 28. PMID 39873544